CLINICAL TRIAL: NCT04966624
Title: Ventilatory Strategy Based on Ultrasound Lung Morphology in Patients With Focal ARDS
Acronym: LUVS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BOUHEMAD Abagri 2021
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Focal Acute Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental)
  Interventions: Procedure: LUVS" ventilatory strategy composed of a bundle of measures
- control (Active Comparator)
  Interventions: Procedure: Ventilatory management according to international recommendations (Société de Réanimation de la Langue Française)

INTERVENTIONS:
Procedure: LUVS" ventilatory strategy composed of a bundle of measures — Ventilation in APRV mode early prone sessions, adjustment of positive expiratory pressure according to the patient's BMI and no curarization
  Arms: interventional
Procedure: Ventilatory management according to international recommendations (Société de Réanimation de la Langue Française) — Ventilatory management according to international recommendations (Société de Réanimation de la Langue Française)
  Arms: control

SUMMARY:
ARDS is characterized by a diffuse, bilateral, extensive alveolar-interstitial infiltrate related to damage to the alveolar membrane.

Studies of lung morphology assessed by CT scan have shown 2 types of ARDS. When the loss of ventilation is posterior and caudal, and the pulmonary parenchyma is otherwise "healthy", ARDS is said to be focal. When the loss of ventilation is diffuse, associated with excess tissue affecting the entire lung parenchyma, ARDS is said to be non-focal or diffuse.

Only one recent multicenter study has evaluated whether individualized PEEP adjustment according to lung morphology (focal vs. non-focal) could improve ARDS survival outcomes compared with standard of care. Results for the primary endpoint, 90-day mortality, were negative. But lung morphology was misclassified on CT occurred 85 (21%) of 400 patients. In addition, per-protocol analysis in which misclassified patients were excluded showed that mortality was significantly lower in the personalized ventilation group than in the control group.

Lung ultrasound may be the ideal bedside imaging technique. The loss of pulmonary aeration and its variations induced by therapeutic maneuvers can be quantified by lung ultrasound. Lung ultrasound is a non-invasive, non-ionizing radiation method that can be easily used at the bedside.

APRV ventilation coupled with spontaneous breathing activity prevents atelectasis formation, recruits less ventilated areas, prevents mechanical ventilation-induced lung injury and improves lung compliance.

The hypothesis is that a "LUVS" ventilatory strategy composed of a bundle of measures all aiming at reopening the atelectatic pulmonary zones in focal ARDS (synergistic effect of spontaneous ventilation in APRV mode, early prone sessions, and adjustment of PEEP according to the patient's BMI), could decrease the number of days under mechanical ventilation, compared to protective ventilation with low tidal volume according to the current international recommendations

ELIGIBILITY:
Inclusion Criteria:

* person who has given oral consent or has been included in an emergency
* Older than 18 years
* On mechanical ventilation for less than 24 hours
* Diagnosis of ARDS for less than 24 hours. ARDS according to the Berlin classification: i.e. arterial oxygen pressure to inspired oxygen fraction ratio less than or equal to 300, with a PEEP greater than or equal to 5, presence of bilateral radiological infiltrates not fully explained by heart failure or volume overload
* Focal ARDS determined on pulmonary ultrasound

Exclusion Criteria:

* person who is not a beneficiary of national health insurance
* person who is subject to a legal measure of protection (curatorship, guardianship)
* pregnant or breastfeeding women
* minor
* Patient having benefited from an invasive mechanical ventilation of more than one week in the previous month;
* ARDS in the previous month;
* Chronic respiratory failure under NIV or long term oxygen;
* Severe acute asthma;
* Lobectomy;
* Pneumothorax;
* Pneumomediastinum;
* Pulmonary fibrosis;
* Morbid obesity with a BMI above 40 ;
* Cancer with metastasis;
* Bone marrow transplantation;
* Chemotherapy-induced neutropenia;
* Cirrhosis with a Child-Pugh score of C;
* Suspected or confirmed intracranial hypertension;
* Concurrent participation in another ARDS study;
* Extensive burns on the torso.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of days without invasive ventilation | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France